CLINICAL TRIAL: NCT01751256
Title: Levobupivacaine Continuous Wound Infiltration and Optimal Standard Analgesia Versus Optimal Standard Analgesia Alone After Cesarean Section.
Brief Title: Additional Effect of Wound Infiltration After Cesarean Section With Optimal Standard Analgesia
Acronym: KTcesar
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Poissy-Saint Germain Hospital (Other)
Responsible Party: Principal Investigator, Claude JOLLY, MD, Poissy-Saint Germain Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PoissyStGermainH
Record Dates: First submitted 2012-12-13; First posted 2012-12-17 (Estimated); Last update posted 2012-12-17 (Estimated); Status verified 2012-12

CONDITIONS: Postoperative Pain; Anesthesia, Local; Breast Feeding
Keywords: Postcesarean Section; Postoperative Pain; Care, Postoperative; Anesthesia, Local; Breast Feeding; Morphine; Pain Measurement; levobupivacaine
MeSH Terms: conditions — Pain, Postoperative; Breast Feeding

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Continuous wound infiltration (Experimental): Subfascial continuous wound infiltration with Levobupivacaine: bolus 50mg and 6.25mg/h for 48 hours through a multiperforated catheter, in addition to Celecoxib 200mg twice a day, paracetamol 1g four times a day, Nefopam 20mg four times a day, and intravenous morphine for 24 hours with Patient Controlled Analgesia pump (1.2mg by bolus, 7 minutes lockout period).
  Interventions: Device: Continuous wound infiltration
- Control (No Intervention): Celecoxib 200mg twice a day, paracetamol 1g four times a day, Nefopam 20mg four times a day, and intravenous morphine for 24 hours with Patient Controlled Analgesia pump (1.2mg by bolus, 7 minutes lockout period).

INTERVENTIONS:
Device: Continuous wound infiltration — Subfascial continuous wound infiltration with Levobupivacaine: bolus 50mg and 6.25mg/h for 48 hours through a multiperforated catheter, in addition to Celecoxib 200mg twice a day, paracetamol 1g four times a day, Nefopam 20mg four times a day, and intravenous morphine for 24 hours with Patient Controlled Analgesia pump (1.2mg by bolus, 7 minutes lockout period).
  Arms: Continuous wound infiltration

SUMMARY:
The purpose of this study is to determine wether wound infiltration brings additional analgesia effect after cesarean section with optimal standard postoperative analgesia

DETAILED DESCRIPTION:
Continuous wound infiltration with local anaesthetic has been shown as a safe and opioid-sparing analgesic method after caesarean section with minimal standard analgesia. We aim to evaluate if this benefit remains when an optimal analgesia is used.

Primary outcome is morphine consumption. Secondary outcomes is pain scores, maternal recovery including breastfeeding, side effects of morphine, nurse workload and maternal satisfaction.

Patients scheduled for caesarean delivery will be eligible for the study.

Patients with emergency caesarean delivery, contraindication to analgesic drugs, hemostasis disorder, ongoing infection, diabetes treated with insulin or chronic opioid use will be excluded from the study.

One group will receive standard analgesia including celecoxib and intravenous morphine for 24 hours with Patient Controlled Analgesia pump. The other group will receive the same standard analgesia with additional levobupivacaine initial bolus followed by a continuous subfascial infiltration of 1.25 mg/ml at 5 ml/h for 48 hours through a multiperforated catheter connected to an elastomeric pump.

Total morphine consumption, pain and any associated complications will be recorded for 72 hours. Women wil be asked to fulfill a questionnaire on the second day after cesarean section, assessing recovery, satisfaction and breastfeeding comfort.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled cesarean section

Exclusion Criteria:

* Emergency cesarean section
* Contraindication to opioids, paracetamol, or local anaesthetic
* Ongoing infection
* Coagulation disorders
* Diabetes treated with insulin
* Chronic opioid use

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2010-06; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Postoperative morphine consumption | 24 first hours after cesarean section
  Quantity of morphine injected by the patient controlled analgesia pump

SECONDARY OUTCOMES:
Pain at mobilization | 4, 8, 12, 16, 20, 24, 36, 48 and 78 hours after skin closure, entrance and exit from the recovery room
  Numerical pain scale during mobilization
Early walking | in the 72 first hours after skin closure
  Time taken for early walking
Resumption of gastrointestinal function | First 72 hours after skin closure
  Interval from the end of surgery until the first gas from the intestinal tract
Treatment tolerance | First 72 hours after skin closure
  Nausea, vomiting, pruritus, excessive sedation
Maternal satisfaction | 2 days after skin closure
  Analogic numerical scale on a specific form
Health staff workload | For the 48 first hours after skin closure
  Number of intervention for nursing, breastfeeding help, and cesarean wound dressing change
Wound infections | the first 10 days after skin closure
  Number of wound infection needing specific cares appeared during the observation time
Local anaesthetic systemic toxicity | During the first 48 hours after skin closure
  Every adverse effect attributed to local anaesthetic by an skilled anesthesiologist
Discomfort due to material | At catheter retrieval
  Discomfort caused by the material and pain at retrieval of the catheter, assessed by an analogic scale on a specific form
Technical problems related to the catheter | During the 48 first hours after skin closure
  Premature withdrawal or occlusion of the catheter
Pain at rest | 4, 8, 12, 16, 20, 24, 36, 48 and 78 hours after skin closure, entrance and exit from the recovery room
  Numerical pain scale at rest
Comfort with Breast Feeding | For the the 48 first hours after skin closure
  Analogic numerical scale on a specific form
All cause morbidity | For the first 10 days after skin closure
  Postpartum hemorrhage or every adverse event occurred during the observation period.

CONTACTS AND LOCATIONS:
Overall Officials: Claude JOLLY, MD, Principal Investigator — Poissy-Saint Germain Hospital
Locations (1):
- Poissy Saint Germain en Laye Hospital, Poissy, France